CLINICAL TRIAL: NCT06338488
Title: The Effectiveness of Dry Needling Treatment in Patients With Shoulder Myofascial Pain Syndrome: Double-blind Randomized Sham-controlled Study.
Brief Title: The Effectiveness of Dry Needling Treatment in Patients With Shoulder Myofascial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hasan Hüseyin Gökpınar, Assistant Professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KutahyaHSU-DRYNEEDLE-SHOULDER
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Prospective double-blind randomized sham-controlled study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In the dry needling application, patients will be blinded to the groups they are randomized into. The evaluator will also be unaware of which group the patients belong to. The practitioner will perform the procedures in both groups using ultrasound guidance, targeting the standard trigger points in the painful shoulder's trapezius and infraspinatus muscles in the study group, and targeting subcutaneous fatty tissue in the same regions in the sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry needling group (study group) (Active Comparator): Real dry needling into the muscle under ultrasound guidance.
  Interventions: Other: Real dry needling
- Sham dry needling group (control group) (Sham Comparator): Sham dry needling into the subcutaneous fatty tissue under ultrasound guidance.
  Interventions: Other: Sham dry needling

INTERVENTIONS:
Other: Real dry needling — dry needling into the muscle under ultrasound guidance.
  Arms: Dry needling group (study group)
Other: Sham dry needling — dry needling into the subcutaneous fatty tissue under ultrasound guidance.
  Arms: Sham dry needling group (control group)

SUMMARY:
Myofascial pain can be diagnosed by the presence of one or more myofascial trigger points (MTrPs), defined as hyperirritable spots in taut bands of skeletal muscle fibers palpable by hand. The treatment of myofascial pain primarily relies on the inactivation of MTrPs, often through manual pressure techniques or dry needling. In manual pressure techniques, the physiotherapist applies increasing pressure directly to the MTrP. In dry needling, acupuncture-like filiform needles are applied to the same point. There are two types of dry needling: superficial dry needling, which penetrates only the skin and superficial muscle, and deep dry needling, which involves inserting a needle directly into the MTrP. The sole or adjunct effectiveness of dry needling treatment targeting the trapezius and infraspinatus muscles has been investigated, particularly in patients with shoulder myofascial pain syndrome. In the study we are planning, a double-blinded efficacy trial will be conducted in patients with shoulder myofascial pain syndrome, where real and sham dry needling applications will be performed under ultrasound guidance, with both the patient and the evaluator blinded. This study design has the potential to make a significant contribution to the literature in this field.

DETAILED DESCRIPTION:
It is planned to enroll 50 patients aged between 18 and 80 years who have been diagnosed with Shoulder Myofascial Pain Syndrome into the study. After signing informed consent forms, eligible patients will be randomized into two different groups using a random number table (randomizer.org) according to inclusion and exclusion criteria. In the study, neither the patient nor the evaluator will know which group they are in; only the physician administering the dry needling treatment will be aware. At the beginning of the study, during weekly follow-ups, and at the end of the study, non-interventional assessment tests will be conducted. Minimal intervention, drug-free dry needling treatment will be administered to patients twice in total, once a week, each session lasting approximately 10-20 minutes with ultrasonographic guidance. Throughout the study period, all patients in both groups will be instructed in detail on the daily exercises they need to perform (trapezius stretching and infraspinatus stretching exercises), as well as on important considerations (avoiding prolonged static positions, etc.). They will be encouraged to perform these exercises daily and mark their completion. Additionally, they will be informed about the selection and usage of medications (only paracetamol) that they can use when necessary, along with instructions on adherence and marking on the provided follow-up form. The entire process will be monitored weekly through the follow-up form provided to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with Shoulder Myofascial Pain Syndrome associated with Infraspinatus trigger point.
* Having a shoulder pain Visual Analog Scale (VAS) score of 6 or higher.
* Ability to read and write

Exclusion Criteria:

* History of shoulder surgery and frozen shoulder syndrome.
* Lesions, atrophy, or scars in the skin around the shoulder.
* Having undergone physiotherapy targeting the shoulder in the last 6 months.
* Undergoing an interventional procedure for shoulder pain in the last 3 months.
* Having used steroids in the last 1 month.
* Special conditions such as epilepsy, pregnancy, injection phobia, etc.
* Inability to comply with the restriction on the use of steroid and non-steroidal anti-inflammatory drugs during the treatment period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: One week after the last intervention, Time frame 4: One month after the last intervention
  "Visual Analog Scale (VAS)" is a measurement instrument often used in healthcare to assess the intensity or characteristics of subjective experiences such as pain. It typically consists of a straight line, usually 10 centimeters in length, with endpoints representing extremes (e.g., "no pain" to "worst imaginable pain"). Patients mark on the line to indicate their subjective experience, and the distance from one endpoint provides a numerical score representing the intensity of the sensation being measured. The VAS is commonly employed in pain assessment but can also be adapted for various other subjective evaluations.
Patient-Specific Functional Scale | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: One week after the last intervention, Time frame 4: One month after the last intervention
  "Patient-Specific Functional Scale" (PSFS). The PSFS is a self-report outcome measure commonly used in healthcare, particularly in physical therapy and rehabilitation settings. It is designed to assess the patient's perceived difficulty in performing specific activities that are relevant to their daily life and function. Identification of Activities: The patient is asked to identify and list three to five activities that they find challenging or have difficulty performing due to their condition or symptoms. Rating Scale: For each identified activity, the patient is asked to rate their current level of difficulty on a numerical scale, often ranging from 0 to 10. A score of 0 indicates no difficulty, while 10 indicates the maximum difficulty. Follow-up Assessments: The same activities and rating scale are used in follow-up assessments to track changes over time or in response to interventions.
Pressure Pain Threshold Measurement | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: Up to 24 hour before the second intervention, Time frame 3: One week after the last intervention, Time frame 4: One month after the last intervention
  "Pressure Pain Threshold Measurement" refers to the assessment of the amount of pressure applied to a specific point on the body before the individual perceives it as painful. This measurement is commonly used in clinical settings to evaluate pain sensitivity and threshold. The process involves gradually applying pressure to a specific area until the individual signals that they begin to feel pain. It is a quantitative way to assess pain perception and is often utilized in research, physical therapy, and other healthcare disciplines to understand pain levels and responses.

SECONDARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention, Time frame 3: One month after the last intervention
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability. Overall total scores range from 0 to 130 with a percentage score of 0 indicating less shoulder disability and 100 indicating more shoulder dysfunction.
The Quick DASH Outcome Measure | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention, Time frame 3: One month after the last intervention
  The Quick DASH is an 11-item measure of the magnitude of disability and symptoms specific to the upper extremity. What is the highest score on QuickDASH? To calculate a QuickDASH score, at least 10 of the 11 items must be completed. Similar to the DASH, each item has 5 response options and, from the item scores, scale scores are calculated, ranging from 0 (no disability) to 100 (most severe disability).
The 12-item Short-Form Health Survey version 2 (SF-12v2) | Time frame 1: Up to 24 hour before the first intervention, Time frame 2: One week after the last intervention, Time frame 3: One month after the last intervention
  The SF-12v2 is a health-related quality-of-life questionnaire consisting of twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). What is the maximum score for SF-12? Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning

CONTACTS AND LOCATIONS:
Overall Officials: Hasan H Gökpınar, Ass. Prof., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University, Kütahya, Türkiye, Turkey (Türkiye)